CLINICAL TRIAL: NCT01704209
Title: Pilot Study of Autologous Fibroblast Injection for Acne Scars, Forehead Lines, Lip Lines, Horizontal Neck Lines, and Static Crow's Feet
Brief Title: Collagen Injections for the Treatment of Acne Scars and Wrinkles
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company stopped making product for cosmetic use. All consented subjects withdrew before any study interventions were performed.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STU67333
Record Dates: First submitted 2012-09-27; First posted 2012-10-11 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Acne Scars; Wrinkles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibroblast Treatment (Experimental): The fibroblast treatment will be randomly injected into one side of the face.
  Interventions: Drug: Fibroblast Treatment
- Vehicle (Placebo Comparator): The vehicle will be injected randomly to the other side of the face.
  Interventions: Procedure: Vehicle

INTERVENTIONS:
Drug: Fibroblast Treatment
  Arms: Fibroblast Treatment
Procedure: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to find out if autologous (your own) fibroblast injections are effective for the treatment of acne scars and wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Bilateral acne scars or have moderate to severe wrinkles
* Subjects in good health
* Subjects has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or lactation
* recent Accutane use in the past 6 months
* prone to hypertrophic and keloidal scarring
* have excessively redundant skin in the treatment area or wrinkles longer than 20 cm total
* have a history of autoimmune disorders, organ transplantation, cancer not in remission, active or chronic skin disease
* have a history of basal-cell carcinoma
* have previously received autologous fibroblast treatment
* have undergone any confounding therapy in the lower two-thirds of the face within 1 year or any investigational treatment within 30 days.
* have an allergy to collagen, bovine products, local anesthetics, gentamicin, or amphotericin B
* subjects who are unable to understand the protocol or to give informed consent
* subjects with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of rater's comparisons at 6 months | Basline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States